CLINICAL TRIAL: NCT05237986
Title: Investigation of the Cognitive Aftereffects of Neurotoxicity in Children and Young Adults With Relapsed/Refractory Hematologic Malignancies Who Receive CAR T-cell Therapy
Brief Title: Cognitive Aftereffects of Neurotoxicity in Children and Young Adults With Relapsed/Refractory Hematologic Malignancies Who Receive CAR T-cell Therapy
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000631; 000631-C
Record Dates: First submitted 2022-02-09; First posted 2022-02-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-12

CONDITIONS: Lymphoma; Leukemia
Keywords: Cogstate; Memory; Leukemia; Lymphoma; Natural History
MeSH Terms: conditions — Lymphoma; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants with relapsed/refractory leukemias or lymphomas, scheduled to receive CAR T-cell therapy.
- Cohort 2: Caregivers (informants)

SUMMARY:
Background:

CAR T-cell therapy is a promising new treatment for blood cancers. During treatment, a person s T-cells are genetically changed to kill cancer cells. Researchers want to learn more about the effects of potential problems that may be associated with this treatment. We are specifically interested in learning if and how this treatment may affect the brain or your thinking skills.

Objective:

To learn if CAR T-cell therapy can affect how children and adults think, process, and remember things.

Eligibility:

People aged 5-35 who have blood cancer that has not responded to treatment, or the blood cancer has come back after treatment, and who will receive CAR T-cell therapy. Caregivers are also needed. All participants must be able to speak and read in English or Spanish.

Design:

Participants will be screened with a medical history.

Information from participants medical records will be collected.

Participants will take tests at home or at NIH to see how well they think, read, learn, remember, reason, and pay attention. The tests will be both computerized and paper/pencil. They will take less than 1 hour to complete.

Participants and a parent/adult observer will complete a 5-minute Background Information Form and a checklist of nervous system symptoms.

If participants are 5 years or older, they will participate in activities to test their ability to do different thinking tasks, like answer questions, complete puzzle patterns, and remember things.

Participants and their caregivers will complete questions to see if they are having specific symptoms related to receiving CAR T-cells. The questions will assess their well-being and needs. The questions will take less than 1 hour to complete.

Some tests and questions will be repeated at different time points in the study.

Participation will last for up to 3 years....

DETAILED DESCRIPTION:
Background:

* Chimeric antigen receptor (CAR) T-cell immunotherapy has rapidly emerged as a successful and breakthrough treatment in pediatric and adult hematologic malignancies. However, significant toxicities can complicate the therapeutic successes of such therapy, including neurologic toxicity associated with cytokine release syndrome (CRS).
* There is a critical need to characterize the subacute and long-term neurocognitive outcomes of participants undergoing CAR T-cell therapies and to compare the results across trials, some of which are first-in-human studies. It is unknown how acute toxicity affects attention, learning, memory, processing speed, and higher order cognition in participants who are cured of their cancer and survive for many years. Information about subacute and long-term neurocognitive sequelae would help determine whether the acute toxicity of specific CAR T-cell therapies needs to be treated and prevented aggressively or whether it is fully reversible without specific intervention.

Objective:

-To evaluate changes in working memory in children and young adults with relapsed/refractory leukemia or lymphoma at 12 months post CAR T-cell therapy

Eligibility:

* Children and young adults (age >= 5 and <=35 years old) with relapsed/refractory leukemias or lymphomas scheduled to have CAR T-cell therapy and their caregivers (informants).
* Participants who can speak and read in English or Spanish

Design:

* This is a multi-center pilot trial to study the neurocognitive effects of CAR T-cell therapy.
* Eligible participants will be seen in one of the enrolling sites.
* Neurocognitive evaluations will be conducted using a computerized test battery (Cogstate) and other paper/pencil tests that assess cognitive processes known to be most affected in participants treated for leukemia or lymphomas as well as patient-reported and observer-reported outcome measures. Participants with the disease and their informants will be enrolled in this study during the preparation of participants for CAR T-cell therapy and followed for up to 3 years post CAR infusion.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants with disease

  * Participants are diagnosed with relapsed/refractory leukemias or lymphomas, and are scheduled to receive CAR T-cell treatment in one of the enrolling sites
  * For participants enrolled on a CAR T-cell treatment protocol, data sharing for the purposes of this study must be allowed.
  * Age >= 5 and <=35 years old
  * Participant must have an eligible caregiver (informant) who is willing to complete assessments about the participant of this study
  * Participants (<18 years, or >=18 years if needed) must have an eligible caregiver to assist with setting up an appropriate test environment for the remote evaluations
  * Participant must be able to speak and understand English or Spanish
  * Participants must have access to a computer or tablet with a camera and an internet connection
  * Participant or parent/guardian must be able to understand and willing to sign a written consent document
* Caregivers (informants)

  * Participants must be able to speak and read in English or Spanish
  * Participants who are caregivers for participants with disease addressed above
  * Age >= 18 years old
  * Participants must have access to a computer or tablet
  * Participants (of children <18 years, or >18 years if needed) must be willing to help set up an appropriate test environment for the remote evaluations
  * Participant is able to understand and willing to sign a written consent document

EXCLUSION CRITERIA:

-Participants with disease who have a pre-existing global intellectual disability (e.g., Down Syndrome)

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with relapsed/refractory leukemias or lymphomas, scheduled to receive CAR T-cell therapy and their caregiver(s).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate changes in working memory in children and young adults with relapsed/refractory leukemia or lymphoma at 12 months post CAR T-cell therapy | 12 months post CAR T-cell therapy
  The changes in working memory (as measured by Cogstate One-Back reaction time standardized score) from baseline to 12-month post-infusion will be determined for each participant and the paired difference will be tested for a change from zero using a paired t-test. If the paired difference is not consistent with a normal distribution, then a Wilcoxon signed rank test may be used instead.

SECONDARY OUTCOMES:
To evaluate changes in additional neurocognitive domains in children and young adults with relapsed/refractory leukemia or lymphoma at 12 months post CAR T-cell therapy | 12 months post CAR T-cell therapy
  The changes in neurocognitive outcomes (reaction time, visual attention, learning and memory, working memory, and executive function) and daily functioning (everyday executive functioning, adaptive behavior, physical and mental health symptoms) from baseline to 12-month post-infusion will be determined for each participant and the paired difference will be tested for a change from zero using a paired t-test. If the paired difference is not consistent with a normal distribution, then a Wilcoxon signed rank test may be used instead.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Wolters, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Children s Hospital of Los Angeles, Los Angeles, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Seattle Children s Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000631-C.html